CLINICAL TRIAL: NCT06103604
Title: The Diagnostic Accuracy and Precision of the Latest Generation Tympanic Thermometers in the Adult and Paediatric Population: Multicentre Cross-sectional Study
Brief Title: Tympanic Thermometers Accuracy
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 507/2023/Oss/IOR
Record Dates: First submitted 2023-10-18; First posted 2023-10-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Fever
Keywords: Thermometers; Sensitivity and Specificity; Hypothermia; Hyperthermia
MeSH Terms: conditions — Fever; Hypersensitivity; Hypothermia; Hyperthermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- in-patients requiring temperature monitoring: The patient at any age whose core temperature is monitored during hospitalisation
  Interventions: Diagnostic Test: latest generation tympanic thermometer

INTERVENTIONS:
Diagnostic Test: latest generation tympanic thermometer — The patient whose core temperature is monitored during hospitalisation has his temperature at tympanic level taken once during the stay. The research nurse will record the core temperature from the monitor on the CRF and, within the next 5 minutes, take the peripheral temperature with the tympanic thermometer three times in a row, recording all three values on the CRF. Subsequently a second operator will always take the temperature 3 times within 5 minutes of the gold standard measurement. Only the first tympanic measurement will then be used to assess accuracy against the gold standard.

SUMMARY:
The aim of the present study is to evaluate the measurement precision and accuracy of the third-generation tympanic thermometer in relation to the measurement modalities considered gold standard. The evaluation of the instrument will be conducted in relation to the different calibration times of the tympanic thermometer, the level of re-training of healthcare personnel in the use of the instrument and the adult and paediatric population subjected to the measurement. Finally, the diagnostic capacity of the instrument in correctly identifying states of hypothermia and febrile elevations will be assessed.

DETAILED DESCRIPTION:
The temperature measurement will be taken on each patient enrolled at a single time by the caregiver for that patient. As the measurements do not depend on which side they are taken, the most convenient side will be chosen. Each patient will only be included once

The research nurse will record the core temperature from the monitor on the CRF and, within the next 5 minutes, take the peripheral temperature with the tympanic thermometer three times in a row, recording all three values on the CRF. Subsequently a second operator will always take the temperature 3 times within 5 minutes of the gold standard measurement. The gold standard (reference tests), as indicated in the literature, can be either the thermometer inserted in the probe placed in the pulmonary artery, or the thermometer inserted in the bladder catheter or oesophageal probe, or directly a rectal thermometer.

Only the first tympanic measurement will then be used to assess accuracy against the gold standard. The other measurements above will only be evaluated for inter and intra reliability. The unit under study is therefore the individual patient at a precise point in time

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients over the age of 4 months
* adults admitted to intensive care and resuscitation
* undergoing surgery who by current practice undergo invasive core temperature measurement

Exclusion Criteria:

* Patients with bilateral auricular inflammatory problems,
* patients who will not use the gold standard for clinical reasons,
* patients or legal guardians who do not consent to participate in the study.

Min Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients admitted to acute hospitals
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Measure of Agreement | The temperature measurement will be taken on each patient enrolled up to 2 weeks
  Measure of Agreement between the thermometer and the gold standard to be assessed by the Bland and Altman method.

SECONDARY OUTCOMES:
accuracy | The temperature measurement will be taken on each patient enrolled up to 2 weeks
  sensitivity, specificity, predictive values, likelihood ratios

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - ASO Azienda Ospedaliera Nazionale SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - Istituto Ortopedico Rizzoli, Bologna
  - Policlinico di S.Orsola Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - Azienda Ospedaliera Universitaria Meyer Istituto di Ricovero e Cura a Carattere Scientifico, Florence
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - APSS Trento, Trento
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona